CLINICAL TRIAL: NCT01470560
Title: Mindfulness-Based Stress Reduction Techniques and Yoga for Treatment of Urinary Urge Incontinence (MBSR-Yoga)
Acronym: MBSR-Yoga
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jan Baker, Advanced Practice Registered Nurse, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00047159
Record Dates: First submitted 2011-11-09; First posted 2011-11-11 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Urinary Incontinence; Urinary Incontinence, Urge
Keywords: Mindfulness; Mindfulness-Based Stress Reduction; Meditation; Yoga
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Urge | interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham Yoga Group Treatment (Sham Comparator): Sham yoga group (control group) will attend 8 weekly sessions for 1-2 hours and will be lead by a certified yoga instructor. The yoga class will be based on Pantajali's Eight Fold Path which is the basis of Yoga. Emphasis will be placed on healthy alignment and ways to pace and adjust poses to make them safe and productive for the body.
  Interventions: Behavioral: Sham Yoga Group
- MBSR Group Treatment (Active Comparator): Mindfulness-Based Stress Reduction (MBSR) was developed by Jon Kabat-Zinn in 1979. MBSR is a group-based intervention, typically provided to up to 30 participants, in a class-based format of eight weekly two hour sessions.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR)

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction (MBSR) — Mindfulness-Based Stress Reduction (MBSR) was developed by Jon Kabat-Zinn in 1979. MBSR is a group-based intervention, typically provided to up to 30 participants, in a class-based format of eight weekly two hour sessions.
  Other Names: MBSR developed by Jon Kabat-Zinn
  Arms: MBSR Group Treatment
Behavioral: Sham Yoga Group — Emphasis will be placed on healthy alignment and ways to pace and adjust poses to make them safe and productive for the body.
  Arms: Sham Yoga Group Treatment

SUMMARY:
Many women experience the accidental loss of urine called urge incontinence or overactive bladder (OAB) incontinence. Women describe this as a sudden, strong desire to pass urine which results in leakage before reaching the toilet. The current usual treatments for urge incontinence include behavioral treatment, physical therapy, and medicines. Although these treatments have been found to be effective in research studies, they are less effective over time in general practice. Because medicines have side effects, many women stop them. The purpose of this study is to explore different treatments that may provide another option for women with urge incontinence that might be effective. This is an initial study to see if these treatments are at least as effective as the usual treatments.

Hypothesis: Does Mind Based Stress Reduction(MBSR)(meditation practices)reduce urinary urge incontinence episodes?

ELIGIBILITY:
Inclusion Criteria:

1. Females at least 18 years of age
2. Five or more urge urinary incontinence episodes on a three-day voiding diary. Urge incontinence episodes will be determined based on voiding diary and subject indication of coincident urge symptoms, allowing self-characterization of incontinence type.
3. Urge predominant (urge >50% of total incontinent episodes) urinary incontinence based on self-reported characterization of incontinent episodes on diary.
4. Request for treatment for urge urinary incontinence.
5. Subject is able to complete all study related items and interviews.

Exclusion Criteria:

1. Any current or recent (past 4 weeks) anticholinergic medication use. Patient may discontinue medication and after 4 weeks may be eligible for study.
2. Past non-pharmacologic treatment for urge incontinence such as supervised behavioral therapy, supervised or unsupervised physical therapy, supervised biofeedback, and transvaginal electrical stimulation.
3. Current symptomatic urinary tract infection that has not resolved prior start of MBSR group.
4. Symptoms of pelvic organ prolapse screened by PFDI (Pelvic Floor Disorder Inventory question #3) "Do you have a bulge or something falling out that you can see or feel in the vaginal area?"
5. Previous or currently implanted neuromodulation (sacral or tibial).
6. Surgically altered detrusor muscle, such as augmentation cystoplasty.
7. Women with known neurologic disease believed to potentially affect urinary function (Multiple sclerosis, spinal cord injuries, myasthenia gravis, Charcot-Marie-Tooth disease).
8. In the opinion of the investigator, inability to understand diary instructions and complete 3-day voiding diary.
9. Subject has been previously diagnosed with interstitial cystitis or chronic pelvic pain syndrome.
10. Currently pregnant or within 6 months postpartum (pregnancy is not excluded for safety reasons but for quality of data)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2011-02; Primary Completion 2012-05 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Pre-Post Leakage Episodes | 0 (Baseline) and 8 weeks
  The primary outcome for the study is the change from baseline in mean number of urge incontinent episodes from pre treatment to post-treatment measured using 3-day voiding diaries.

SECONDARY OUTCOMES:
Quality of Life | 0 (Baseline) and 8 weeks
  Secondary Outcome Measures are a change from baseline in the Overactive Bladder Questionnaire (OABq-SF) scores and proportion of subjects reporting improvement from the Patient Global Impression of Improvement (PGI-I)).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States